CLINICAL TRIAL: NCT02889809
Title: Study HZA114971, A Multicentre Randomised, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Effects of a One-Year Regimen of Orally Inhaled Fluticasone Furoate 50 mcg Once Daily on Growth Velocity in Prepubertal, Paediatric Subjects With Asthma
Brief Title: Effects of a Orally Inhaled Fluticasone Furoate on Growth Velocity in Prepubertal, Paediatric Subjects With Asthma Over a Year
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 114971
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Results first posted 2022-01-04 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-12

CONDITIONS: Asthma
Keywords: Growth Velocity; Prepubertal; Asthma; Paediatric
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate; montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fluticasone furoate 50 mcg (Experimental): During run-in period, subjects will receive inhaled placebo for 16 weeks using ELLIPTA inhaler. Followed by treatment period where subjects will receive inhaled FF 50 mcg administered once daily in the morning for 52 weeks using ELLIPTA inhaler. Subjects will also receive open-label montelukast (4 milligrams [mg] for subjects who are 5 years old and 5 mg for subjects who are >= 6 years old) to be administered as one tablet of montelukast each evening for the duration of the study. Each subject will receive a SABA (albuterol/salbutamol [inhalation aerosol or nebuliser]) to be used as needed throughout the entire study period as rescue medication for symptomatic relief of asthma symptoms.
  Interventions: Drug: Fluticasone furoate; Drug: Placebo; Drug: Montelukast; Drug: Short Acting Beta 2 Agonist
- Placebo (Placebo Comparator): During run-in period, subjects will receive inhaled placebo for 16 weeks using ELLIPTA inhaler. Followed by treatment period where subjects will receive inhaled placebo administered once daily in the morning for 52 weeks using ELLIPTA inhaler. Subjects will also receive open-label montelukast (4 milligrams [mg] for subjects who are 5 years old and 5 mg for subjects who are >=6 years old) to be administered as one tablet of montelukast each evening for the duration of the study. Each subject will receive a SABA (albuterol/salbutamol [inhalation aerosol or nebuliser]) to be used as needed throughout the entire study period as rescue medication for symptomatic relief of asthma symptoms.
  Interventions: Drug: Placebo; Drug: Montelukast; Drug: Short Acting Beta 2 Agonist

INTERVENTIONS:
Drug: Fluticasone furoate — Fluticasone furoate will be supplied as 50 mcg per blister dry white powder for inhalation using ELLIPTA inhaler.
  Arms: Fluticasone furoate 50 mcg
Drug: Placebo — Placebo will be supplied as dry white powder Lactose for inhalation using ELLIPTA inhaler.
Drug: Montelukast — Montelukast will be supplied as 4 mg chewable tablet (5 year old subjects) and as 5 mg chewable tablet (>=6 year old subjects)
Drug: Short Acting Beta 2 Agonist — Albuterol/salbutamol will be supplied as inhalation aerosol or nebulizer.

SUMMARY:
There is a regulatory requirement to evaluate the extent of reduction (if any) of growth velocity associated with inhaled corticosteroid (ICS) containing products that are to be administered to children, and to this end there is Food and Drug Administration (FDA) regulatory guidance. This is a randomised, single-blind (run-in period)/double-blind (treatment period), parallel group, placebo controlled, multicentre study to assess the effect of once daily (OD) inhaled fluticasone furoate (FF) 50 microgram (mcg) on growth velocity in prepubertal asthmatic children on a background therapy of open-label montelukast. This study will be conducted over a total duration of approximately 76 weeks: 16-week run-in period (single-blind placebo inhaler), 52-week double-blind treatment period (inhaled FF 50 mcg /placebo administered OD in the morning for 52 weeks) and 8-week follow-up period. The purpose of the study is to evaluate the magnitude of effect (with a level of precision) on growth velocity of prepubertal asthmatic paediatric subjects (aged 5 to <9 years) following administration of OD inhaled FF 50 mcg for one year. This study fulfills European Union (EU) and United States (US) regulatory requirements for the evaluation of potential growth suppression in children.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects.
* Age: Males between 5 and <9 years old; Females between 5 and <8 years old.
* Subjects must be pre-pubertal (Tanner Stage 1).
* Height centile between 3% and 97% based on local growth charts.
* Subjects with body weight and body mass index that is between 3rd and 97th centile based on the United State (US) Centres for Disease Control and Prevention (CDC) standard statistics or any local standards outside the US.
* A documented history of symptoms consistent with a diagnosis of asthma for at least 6 months prior to Visit 1.
* A pre-bronchodilatory forced expiratory flow in 1 second (FEV1) at Visit 1 (Screening) of between >=60% to <=95% predicted. There should be no short acting beta 2 agonist (SABA) use within 4 hours of this measurement.
* Able to replace their current SABA treatment with study supplied rescue albuterol/salbutamol provided at Visit 1 for use as needed for the duration of the study.
* A childhood asthma control test (cACT) score of >19.
* Subjects should have required at least one course of corticosteroid for their asthma (inhaled or oral) in the past year.
* There must be no ICS use within 6 weeks of Visit 1 (Screening).
* There must be no oral corticosteroids use within 12 weeks of Visit 1 (Screening).
* Using one or more of the following asthma therapies prior to entry into the study:

Short acting beta-agonist (SABA) inhaler alone (example given [e.g.] salbutamol) on an as needed basis and/or regular non-ICS controller medications for asthma (e.g. cromones or leukotriene receptor antagonists).

- Written informed consent from at least one parent/care giver (legal guardian) and accompanying informed assent from the subject (where the subject is able to provide assent) prior to admission to the study. If applicable, subject must be able and willing to give assent to take part in the study according to local requirement. The study investigator is accountable for determining a child's capacity to assent for participation in a research study, taking into consideration any standards set by the responsible Independent Ethics Committee (IEC). Subject and their legal guardian(s) understand that they must comply with study medication administration regimens and study assessments including recording of symptom scores and rescue albuterol/salbutamol use, attending all study visits, and being accessible by telephone.

Exclusion Criteria:

* Growth Criteria: Any previous or current condition that affects growth, including sleep disorders, endocrine disorders, skeletal dysplasia, Turner and Noonan syndromes, Marfan, Beckwith-Wiedeman and Sotos syndromes, Klinefelter's syndrome, coeliac disease, inflammatory bowel diseases and renal failure or any significant abnormality or medical condition that is identified at the screening medical assessment (including serious psychological disorder) that is likely to interfere with the conduct of the study.
* Subjects with premature adrenarche.
* A child who is unable to stand, or who finds standing difficult due to illness or physical disabilities should be excluded.
* Disease Criteria: Subjects with a history of asthma exacerbation requiring the use of systemic corticosteroids (tablets, suspension, or injection) for at least 3 days or use of a depot corticosteroid injection within 3 months or those requiring hospitalisation for asthma (within 6 months) prior to screening.
* Culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear that is not resolved within 4 weeks of Visit 1 and led to a change in asthma management or, in the opinion of the Investigator, is expected to affect the subject's asthma status or the subject's ability to participate in the study.
* Clinical visual evidence of candidiasis at Visit 1 (Screening).
* Any significant abnormality or medical condition identified at the screening medical assessment that in the Investigator's opinion, preclude entry into the study due to risk to the subject or that may interfere with the outcome of the study.
* General: Prior use of any medication or treatment that might affect growth including, but not limited to: amphetamines, anticonvulsants, biphosphonates, calcitonin, calcitriol, erythropoietin, growth hormone, methylphenidate, phosphate binders, antithyroid drugs (e.g., Methimazole) or thyroid hormone.
* Use of any of the prohibited medications listed in the study protocol.
* Hypersensitivity: Known hypersensitivity to corticosteroids, leukotrienes, or any excipients in the ELLIPTA (ELLIPTA is a Glaxosmithkline owned trademark for dry powder inhaler) inhaler and study tablets.
* Milk Protein Allergy: History of severe milk protein allergy.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than 4 investigational medicinal products within 12 months prior to the first dosing day.
* Children who are an immediate family member of the participating Investigator, sub-Investigator, study coordinator, or employee of the participating Investigator.
* The Parent or Guardian has a history of known or suspected psychiatric disease, intellectual deficiency, substance abuse or other condition (e.g. inability to read, comprehend or write) which may affect: validity of consent to participate in the study; adequate supervision of the subject during the study; compliance of subject with study medication and study procedures (e.g. completion of daily diary, attending scheduled clinic visits); subject safety and well-being.
* Children in care: Children who are wards of the government or state are not eligible for participation in this study.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 477 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (40):
- United States (15):
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Homestead, Florida
  - GSK Investigational Site, Loxahatchee Groves, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Gainesville, Georgia
  - GSK Investigational Site, Ypsilanti, Michigan
  - GSK Investigational Site, Bellevue, Nebraska
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Waco, Texas
- Argentina (4):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Lanús, Buenos Aires
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
- Poland (8):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Gdansk-Wrzeszcz
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Skarżysko-Kamienna
  - GSK Investigational Site, Szczecin
  - GSK Investigational Site, Tarnów
- Romania (4):
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, ClujNapoca
  - GSK Investigational Site, Sangiorgiu de Mures
- Russia (6):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Voronezh
  - GSK Investigational Site, Yaroslavl
- South Africa (3):
  - GSK Investigational Site, Middelburg, Mpumalanga
  - GSK Investigational Site, Bellville
  - GSK Investigational Site, Cape Town

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency

REFERENCES:
- [Background] Bareille P, Imber V, Crawford J, Majorek-Olechowska B, Karam-Absi Z, Stone S, Birk R. A multicenter randomized, double-blind, placebo-controlled, parallel-group study to evaluate the effects of a 1-year regimen of orally inhaled fluticasone furoate 50 microg once daily on growth velocity in prepubertal, pediatric participants with well-controlled asthma. Pediatr Pulmonol. 2023 Dec;58(12):3487-3497. doi: 10.1002/ppul.26679. Epub 2023 Sep 20. PMID 37728224

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter, randomized, double-blind, placebo-controlled study to evaluate the effects of a one-year regimen of orally inhaled fluticasone furoate (FF) 50 micrograms (mcg) once daily on growth velocity in prepubertal, pediatric participants with asthma.
Pre-assignment Details: Total 477 participants were enrolled in this study.
Groups:
- Placebo: Participants received a single-blind placebo inhaler during a 16-week run-in period. After run-in period inhaled placebo was administered once daily (OD) in the morning for 52 weeks during the double-blind treatment period. Participants also received open-label montelukast one tablet orally in the evening (4 milligrams [mg] for participants who were 5 years old and 5 mg for participants who were greater than or equal to [>=] 6 years old) as background therapy from the run-in period through to the end of follow-up (8 weeks) period.
- FF 50 mcg: Participants received received a single-blind placebo inhaler during a 16-week run-in period. After run-in period inhaled FF 50 mcg was administered via ELLIPTA inhaler once daily in the morning for 52 weeks during double-blind treatment period. Participants also received open-label montelukast one tablet orally in the evening (4 mg for participants who were 5 years old and 5 mg for participants who were >=6 years old) as background therapy from the run-in period through to the end of follow-up (8 weeks) period.
Period: Overall Study
Arm/Group | Placebo | FF 50 mcg
Started | 239 | 238
Completed | 196 | 205
Not Completed | 43 | 33
Not completed — Withdrawal by Subject | 30 | 21
Not completed — Lost to Follow-up | 1 | 1
Not completed — Site Closed | 12 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | FF 50 mcg | Total
Number analyzed (Participants) | 239 | 238 | 477
Age, Continuous [Mean (Standard Deviation); unit: Years] | 6.1 (1.07) | 6.3 (1.02) | 6.2 (1.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 94 | 178
  Male | 155 | 144 | 299
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 13 | 13 | 26
  Asian - Central/South Asian Heritage | 0 | 1 | 1
  Multiple | 18 | 20 | 38
  White - Arabic/North African Heritage | 3 | 3 | 6
  White - Mixed Race | 1 | 0 | 1
  White - White/Caucasian/European Heritage | 204 | 201 | 405

OUTCOME MEASURES:

1. Primary Outcome: Growth Velocity (Centimeter Per Year) Over the Double-blind Treatment Period, as Determined by Stadiometry
Description: Three reproducible height measurements were taken using a stadiometer at each visit and were recorded to nearest 1/10th of centimeter. Each set of triplicate measurements was averaged to derive one estimated height per participant per visit. Growth velocity was calculated for each participant over double-blind treatment period (up to 52 weeks [wk]) by fitting a regression line to averaged height measurements at each visit for that participant during period. Slope of this regression line was participant's growth velocity for double-blind treatment period. Treatment policy estimand was assessed, including all on- and post-treatment data. Baseline was included as covariate which was calculated based on stadiometric height measurements recorded at Visits 1(wk -16), 3(wk-8), and 5(wk0), data from at least two of these visits were used to fit a simple linear regression line against time and the slope of the fitted regression line was the participant's Baseline growth velocity.
Time Frame: Up to 52 weeks
Population: Growth Population comprised of all Intent to Treat (ITT) participants who have stadiometric height assessments from at least three post-randomization, on-treatment clinic visits (i.e., including all available height measurements after Visit 5 [wk 0] up to and including Visit 18 [wk 52], without exclusion) during the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: Centimeter per year
Arm/Group | Placebo | FF 50 mcg
Number analyzed (Participants) | 226 | 231
Centimeter per year | 6.065 (0.1090) | 5.905 (0.1078)
Statistical Analysis 1: Comparison: Placebo vs FF 50 mcg; Test type: Other; Least Square (LS) Mean Difference = -0.160, 95% CI 2-sided [-0.462 to 0.142] — Analysis was performed using an analysis of covariance (ANCOVA) model adjusting for Baseline growth velocity, age at Visit 1, gender and country

2. Secondary Outcome: Percentage of Participants Below the Third Percentile of Growth Velocity During Double-blind Treatment Period
Description: Three reproducible height measurements were taken using stadiometer at each visit&were recorded to nearest 1/10th of a centimeter.Each set of triplicate measurements was averaged to derive one estimated height per participant per visit.Growth velocity(GV)was calculated for each participant over double-blind treatment(up to 52 weeks)period by fitting regression line to height measurements recorded for that participant during period.Each participant's double-blind(DB) treatment period GV was calculated based on all on &off treatment height data &was programmatically compared to data values from Standards from Birth to Maturity for Height,Weight,Height Velocity, established in British Children(1965)&further updated for North American children(1985)using 3rd percentile value of age closest to participant's age at end of endpoint(i.e.either end of participant's DB treatment period [Visit18 Wk 52]/withdrawal from study[Early Withdrawal Visit]).Percentage values presented is rounded off.
Time Frame: Up to 52 weeks
Population: Growth Population
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | FF 50 mcg
Number analyzed (Participants) | 226 | 231
Percentage of participants | 9 | 7

3. Secondary Outcome: Percentage of Participants With Change in Growth Velocity Quartiles From Baseline to Endpoint
Description: Growth velocity(GV) quartile(defined as 1st quartile(1Q)=1st-25th percentile,2Q=26th-50th percentile,3Q=51st-75th percentile,4Q=76th-100th percentile) was determined at Baseline&endpoint.Endpoint was defined as slope of simple linear regression of average stadiometric height recorded at week 28& upto wk52.Baseline growth velocity was calculated as slope from simple linear regression of average stadiometric height recorded at wk-16,-8&0.Baseline GV was programmatically compared to reference for standard height data using participant's estimated age at wk0& age in reference data closest to actual age of participant to determine Baseline GV quartile.Endpoint GV was programmatically compared to reference data using participant's age at endpoint & age in reference data that was closest to actual age of participant to determine endpoint GV quartile. Any increase/decrease indicates any increase/decrease in quartiles with reference to Baseline. Percentage values presented is rounded off.
Time Frame: Baseline and Endpoint (Week 28[Visit 12] up to and including Week 52 [Visit 18])
Population: Growth Population. Only those participants with data available at the specified data points were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | FF 50 mcg
Number analyzed (Participants) | 216 | 223
Percentage of Participants
  Any increase | 33 | 32
  Any decrease | 34 | 38

4. Secondary Outcome: Growth Velocity Over the First 12 Weeks of Double-blind Treatment Period
Description: Growth velocity was calculated for each participant over double blind period by fitting regression line to height measurements recorded for that participant during period.Slope of this regression line was participant's growth velocity for double-blind treatment period.In order to be included in this analysis,participant must have data from Visit8(Wk 12) stadiometric height assessment.Baseline was included as covariate which was calculated based on stadiometric height measurements recorded at Visits 1(wk -16),3(wk-8),& 5(wk0),data from at least two of these visits were used to fit simple linear regression line against time&slope of fitted regression line was participant's Baseline growth velocity.All available height data collected during double-blind treatment period upto Visit8(Wk12) while participant was on randomized double-blind treatment was considered.ANCOVA model was used to estimate mean treatment difference in growth velocity over 1st 12weeks of double-blind treatment period.
Time Frame: Up to 12 weeks (Visit 8) of double-blind treatment period
Population: Growth Population. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Centimeter per year
Arm/Group | Placebo | FF 50 mcg
Number analyzed (Participants) | 210 | 211
Centimeter per year | 6.222 (0.1845) | 6.281 (0.1841)
Statistical Analysis 1: Comparison: Placebo vs FF 50 mcg; Test type: Other; LS Mean Difference = 0.059, 95% CI 2-sided [-0.455 to 0.572] — Analysis was performed using an ANCOVA model adjusting for Baseline growth velocity, age at Visit 1(wk -16), gender and country

5. Secondary Outcome: Change in Height Standard Deviation Scores (SDS) From Baseline to Endpoint
Description: Each participant's SDS for each of three required stadiometric height measurements was calculated as:(observed height measurement-standard median height for age at Visit [week-16]) divided by (/) ([standard 95th height percentile for age at visit-standard 5th height percentile for age at visit]/[2*1.645]).Standard median, 95th percentile, & 5th percentile values were obtained from standard tables (Guidance for Industry Orally Inhaled & Intranasal Corticosteroid). SDS for each height stadiometric measurement at each visit was calculated using percentiles from standard tables & averaged for each participant before being summarized by treatment group. A reduction in SDS over time indicates growth deceleration & an increase in SDS over time means growth acceleration.Baseline was defined as height SD score at Visit 5 (week 0). Endpoint was defined as height SD score at Visit 18 (week52) (on- & off-treatment data). Change from Baseline was calculated as Endpoint value minus Baseline value.
Time Frame: Baseline (Week 0 [Visit 5]) and up to Endpoint (Week 52 [Visit 18])
Population: Growth Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Standard Deviation Score
Arm/Group | Placebo | FF 50 mcg
Number analyzed (Participants) | 196 | 202
Standard Deviation Score | -0.02 (0.281) | -0.04 (0.281)

6. Secondary Outcome: Number of Participants With Non-serious Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE is defined as any untoward medical occurrence that, at any dose which results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations as per investigator's judgement.
Time Frame: Up to 76 weeks
Population: Intent-to-Treat Population comprised of all randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | FF 50 mcg
Number analyzed (Participants) | 239 | 238
Participants
  Any SAEs | 8 | 6
  Any Non-serious AEs | 105 | 99

7. Secondary Outcome: Number of Participants With On-treatment Asthma Exacerbations Over Double-blind Treatment Period
Description: An exacerbation is defined as deterioration of asthma requiring the use of systemic corticosteroids (tablets, suspension, or injection) for at least 3 days or a single depot corticosteroid injection, or an in-patient hospitalization or emergency department (ED) visit due to asthma that required systemic corticosteroids. Number of participants with on-treatment asthma exacerbations during double-blind treatment period is presented.
Time Frame: Up to 52 weeks
Population: Intent-to-Treat Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | FF 50 mcg
Number analyzed (Participants) | 239 | 238
Participants | 22 | 7

ADVERSE EVENTS:
Time Frame: All cause mortality, non-serious adverse events (AEs) and serious AEs were collected up to 76 weeks
Description: All-cause mortality, non-serious AEs and SAEs were collected in Intent-to-Treat Population which comprised of all randomized participants who received at least one dose of study treatment.
Arm/Group | Placebo | FF 50 mcg
All-Cause Mortality (participants affected / at risk) | 0/239 | 0/238
Serious Adverse Events (participants affected / at risk) | 8/239 | 6/238
Other Adverse Events (participants affected / at risk) | 105/239 | 99/238
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=239) | FF 50 mcg (N=238)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adenoviral haemorrhagic cystitis (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Testicular appendage torsion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=239) | FF 50 mcg (N=238)
Pyrexia (General disorders) | 18 (23) | 13 (15)
Bronchitis (Infections and infestations) | 12 (13) | 9 (11)
Influenza (Infections and infestations) | 7 (8) | 11 (11)
Nasopharyngitis (Infections and infestations) | 25 (31) | 23 (26)
Pharyngitis (Infections and infestations) | 9 (10) | 3 (3)
Respiratory tract infection viral (Infections and infestations) | 4 (7) | 10 (11)
Rhinitis (Infections and infestations) | 18 (26) | 16 (18)
Upper respiratory tract infection (Infections and infestations) | 33 (57) | 29 (63)
Headache (Nervous system disorders) | 12 (24) | 10 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (23) | 12 (15)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 8 (9)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial

DOCUMENTS (2):
  • Study Protocol (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/09/NCT02889809/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/09/NCT02889809/SAP_001.pdf